CLINICAL TRIAL: NCT07273773
Title: Evaluation of the Rigicon Infla10® Inflatable Penile Prosthesis (IPP) A Prospective, Multicenter, Single-Arm Performance-Goal Study
Brief Title: Evaluation of the Rigicon Infla10® Inflatable Penile Prosthesis (IPP) for Erectile Dysfunction
Acronym: UNITED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC2025_UNITED
Record Dates: First submitted 2025-11-26; First posted 2025-12-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Erectile Dysfunction (ED)
Keywords: Rigicon; Infla10; inflatable penile prosthesis; penile prosthesis; Dynamic; erectile dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Patients implanted with Infla10® Pulse™ Dynamic Inflatable Penile Prosthesis (Experimental): Male subjects 22 years of age and older who are implanted with an Rigicon Infla 10® Three-Piece Inflatable Penile Prosthesis for erectile dysfunction.
  Interventions: Device: Rigicon Infla10® Inflatable Penile Prosthesis (IPP)

INTERVENTIONS:
Device: Rigicon Infla10® Inflatable Penile Prosthesis (IPP) — Medical Device: Infla10® Pulse™ Dynamic Inflatable Penile Prosthesis
  • Other Names: Inflatable Penile Prosthesis (IPP) Treatment: Erectile dysfunction

SUMMARY:
This study evaluates the long-term safety and effectiveness of the Rigicon Infla10® Inflatable Penile Prosthesis in patients with erectile dysfunction. The study follows patients implanted with the Rigicon Infla10® Pulse™ Dynamic Inflatable Penile Prosthesis for up to 3 years after implantation.

DETAILED DESCRIPTION:
Erectile dysfunction (ED) is a common male sexual dysfunction associated with a reduced quality of life for patients and their partners. Incidence of ED increases with age and is associated with depression, obesity, diabetes mellitus, hypertension, cardiovascular disease and benign prostatic hyperplasia. ED is diagnosed with symptoms of (1) inability to attain or sustain a penile erection during sexual activity and (2) a reduction of penile rigidity in >75% of sexual encounters during six months period. ED is estimated to affect approximately 52% of men in age of 40 to 70 years. It is projected in 2025, the worldwide ED prevalence of about 322 million. ED usually has organic causes, such as damage of arteries, smooth muscle and fibrous tissue. This results in impairment of blood flow to and from penis due to diabetes, renal disease, atherosclerosis and vascular disease.

Management of ED involves lifestyle modification, medical, surgical interventions, and possibly, in the future, tissue- engineering or cellular or gene therapy. Oral phosphodiesterase type 5 inhibitor (PDE5i), which works with sexual stimulation, is an effective medical therapy for ED with an excellent safety profile. Intracavernosal injection or topical application of vasoactive drugs have also been studied. The first inflatable penile prosthesis was introduced in 1973, and current models of inflatable penile prostheses include the AMS 700 series, Coloplast Titan device and Zephyr ZSI device. A patient-activated inflatable penile prosthesis (IPP) provides patients with a means to achieve dependable spontaneity for intercourse.

Rigicon has developed a three-piece inflatable penile prosthesis (IPP) (Infla10®) for the treatment of ED. This study is to assess the safety and effectiveness of the Rigicon IPP in treating ED. Clinical literature and preclinical testing, including biocompatibility, device validation and verification, and animal studies support the safety and efficacy of this device for the intended therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male ≥22 years of age.
2. Diagnosed with erectile dysfunction (impotence).
3. Agree to receive Infla10® three-piece IPP as an ED treatment.
4. Willing to complete all protocol required for follow-up visits and tests.

Exclusion Criteria:

1. Contraindication to general anesthesia.
2. Known allergy or sensitivity to product materials as indicated in the device labeling.
3. Previous penile prosthesis or prior enlargement surgeries
4. Diagnosed penile sensory neuropathy.
5. Patients who are receiving immunosuppressive drugs or have a history of kidney transplantation.
6. Patients who are receiving chemotherapy at the time of enrolment.
7. Diagnosed with fibrotic disease, such as priapism or Peyronie's disease or Chordee.
8. Compromised immune system, such as systemic lupus erythematosus, discoid lupus, or scleroderma.
9. Uncontrolled diabetes (HbA1c ≥ 9.0% [≈75 mmol/mol], measured within 90 days prior to surgery.
10. Bleeding disorder or coagulopathy that may in the judgment of the investigator preclude safe procedure.
11. Active urogenital infection or active skin infection in region of surgery or systemic infection at the time of assessment.
12. Clinically significant comorbidities or presence of unstable conditions (e.g. cardiovascular, lung, renal [serum creatinine > 2.0 mg/dl], hepatic, bleeding disorders, or metabolic impairment) that may confound the results of the study or in the judgment of the physician investigator preclude safe procedure.
13. Lacking manual dexterity or mental abilities necessary to operate the device.
14. Expected life expectancy < two years.
15. Unwilling or unable to sign the Informed Consent.
16. Unwilling or unable to comply with the follow-up study requirements.
17. Psychogenic erectile dysfunction
18. Currently participating in an investigational drug or another investigational device exemption (IDE) study.
19. The cognitively challenged subjects and subjects with any cognitive disorder that interferes with or precludes direct and accurate communication with the study investigator regarding the study or affects the ability to complete the study questionnaires.
20. Incarcerated subjects
21. Subjects who are currently using, or who have not previously attempted and failed, standard non-surgical ED therapies including oral or topical treatments.

Min Age: 22 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 182 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
The primary safety outcome is the proportion of participants free from any device- or procedure-related adverse event of CTCAE Grade ≥2 through 12 months post-procedure, graded per CTCAE v5.0 and IPP-specific mapping. | 12 months
  Success will be concluded if the two-sided 95 percent confidence interval (equivalently, one-sided 97.5 percent) for the 12-month proportion has its lower bound strictly greater than 0.90 as specified in the statistical plan.
The primary effectiveness endpoint is a binary "pass" or "fail" objective axial rigidity test, assessed at 12 months. | 12 months
  The objective axial rigidity test will use a calibrated axial-rigidity device to measure vertical displacement of the fully inflated penis under a standardized 650-gram load. ≤15 mm displacement will be counted as a "pass".
  Success will be concluded if the two-sided 95 percent confidence interval for the 12-month success proportion has its lower bound strictly greater than the pre-specified performance goal in the statistical plan.

SECONDARY OUTCOMES:
Percentage of patients free from revision or explant surgeries at 12 months. | 12 months
  This secondary endpoint will summarize "revision- or explant-free survival" using Kaplan-Meier methods, with participants without an event right-censored at last contact.
International Index of Erectile Function - Erectile Function (IIEF-EF) Domain Score | Baseline (pre-implantation) and Months 3, 6, 12, 18, 24, and 36 post-implantation.
  The Erectile Function (EF) domain of the IIEF-15 questionnaire (Items 1-5 and 15) will be used to assess patient erectile function. Change from baseline in the EF domain total score will be reported at each time point. The questionnaire may be completed remotely via ePRO.
  Scale / Range: 6-30 points Direction: Higher scores indicate better erectile function. Assessment Schedule: Baseline and Months 3, 6, 12, 18, 24, and 36.
Rosenberg Self-Esteem Scale (RSES) Total Score | Baseline (pre-implantation) and Months 3, 6, 12, 18, 24, and 36 post-implantation.
  The 10-item Rosenberg Self-Esteem Scale (RSES) is a validated self-report instrument used to measure global self-worth by assessing positive and negative feelings about the self. The total RSES score will be used as a secondary endpoint to evaluate change in participant self-esteem and psychosocial well-being following device implantation.
  Administration and scoring: Each item is rated on a 4-point Likert scale (1 = Strongly Disagree to 4 = Strongly Agree). Items 2, 5, 6, 8, and 9 are reverse scored. The total score ranges from 10 to 40, with higher scores indicating greater self-esteem.
  Analysis: Change from baseline in total RSES score will be summarized at each time point as mean ± standard deviation with 95% confidence intervals, and formally tested within the pre-specified hierarchical secondary endpoint sequence.
  Scale / Range: 10-40 points Direction: Higher scores indicate higher self-esteem (better outcome).
Adverse Events | 36 months
  Descriptive tabulations by system organ class and preferred term, including device-relatedness and seriousness, and rates for typical post-IPP events categorized as AEs, SAEs, and UADEs.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Perito Urology, Coral Gables, Florida
  - Atlanta Cosmetic Urology, Atlanta, Georgia
  - Dr. Levine Men's Health, Chicago, Illinois
  - Kramer Urology, Hyannis, Massachusetts
  - Premier Medical Group, New Windsor, New York
  - Washington Heights Urology, New York, New York
  - Sun Health Clinic, Arlington, Texas
  - Vitality Urology Institute, Houston, Texas